CLINICAL TRIAL: NCT01639937
Title: Quantitative Myocardial Perfusion, Myocardial Scarring and Their Contribution to Late Clinical Decompensation in Adults With Congenital Heart Disease
Brief Title: Myocardial Perfusion and Scarring in Congenital Heart Disease
Status: Terminated | Type: Observational
Why Stopped: PI is leaving NHLBI, sample size is too small.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Children's National Research Institute (Other); Suburban Hospital (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120158; 12-H-0158
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Congenital Heart Disease
Keywords: Cardiac MRI; Congestive Heart Failure; Cardiac Fibrosis; Late Gadolinium Enhancement
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Subjects with palliated congenital heart disease including, but not limited to, d TGA, ccTGA, single ventricles, hypoplastic left heart syndrome and tricuspid atresia will be recruited

SUMMARY:
Background:

- People with congenital heart disease may develop heart failure earlier that those who do not have the disease. One theory to explain this is that the heart s own blood supply may be different in people with congenital heart disease. Problems with this blood supply can severely damage the heart. This damage can be studied with a heart imaging test called a cardiac magnetic resonance imaging (MRI) scan. Researchers want to use this type of scan to look at the blood supply to the heart in people with congenital heart disease.

Objectives:

- To learn more about the blood supply to the heart in people with congenital heart disease.

Eligibility:

- Individuals at least 18 years of age who have heart defects caused by congenital heart disease.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have a cardiac MRI scan to look at the blood flow to the heart.
* Participants will also have a heart stress test to measure heart function during exercise.
* Other imaging studies of the heart may be performed to collect more information on heart function.

DETAILED DESCRIPTION:
This is a study of the perfusion of the myocardium in adults with specific forms of repaired congenital heart disease using established cardiac MRI techniques and correlating perfusion with clinical outcomes. Our objectives are to examine myocardial perfusion both during stress and at rest in adults with repaired or palliated congenital heart disease as well as quantify ventricular function, regional myocardial strain and evidence of myocardial fibrosis with quantitative measures of myocardial perfusion. The specific aim of this study is to understand whether clinical subendocardial perfusion defects contribute to the late decompensation of adult subjects that have single ventricle physiology and adult subjects that have a systemic right ventricle.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for All Arms of the Protocol:

* Subjects 18 years of age or older
* All defects that have a right ventricle that supports the systemic circulation
* All defects with a functional single ventricle
* Written informed consent

EXCLUSION CRITERIA:

Exclusion Criteria for All Arms of the Protocol:

* Subjects with a contraindication to MRI scanning will be excluded. These contraindications include subjects with the following devices:

  * Central nervous system aneurysm clips
  * Implanted neural stimulator
  * Implanted cardiac pacemaker or defibrillator
  * Cochlear implant
  * Ocular foreign body (e.g. metal shavings)
  * Implanted Insulin pump
  * Metal shrapnel or bullet
* Severe heart damage that makes it difficult to breathe while lying flat
* Pregnant women (Women of childbearing potential who are uncertain as to whether they are pregnant will be required to have a screening urine or blood pregnancy test)
* Subjects with active symptoms of myocardial ischemia occurring despite maximally tolerated doses of oral antianginal therapy and intravenous nitroglycerin

Furthermore, the following subject groups will be excluded from studies involving the administration of MRI contrast agents:

* lactating women unless they are willing to discard breast milk for 24 hours after receiving gadolinium
* renal disease (estimated glomerular filtration rate [eGFR] < 30 ml/min/1.73 m2 body surface area)

The eGFR will be used to estimate renal function if reported by the laboratory. Otherwise, estimated glomerular filtration rate (eGFR) can be based on the Modification of Diet in Renal Disease (MDRD) study equation (see below) in subjects with stable renal function. This formula is not applicable to subjects with acute renal insufficiency:

eGFR (ml/min/1.73 m2) = 175 x (serum creatinine)-1.154 x (age)-0.203 x 0.742 (if the subject is female) x 1.212 (if the subject is black)

Additional Exclusion Criteria for Vasodilator Stress MRI:

* Myocardial infarction within 24 hours
* Uncontrolled heart failure
* Uncontrolled asthma or emphysema
* Ventricular arrhythmia (sustained ventricular arrhythmia at the time of MR scan)
* Second degree heart block or higher

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled at the NIH Clinical Center, Suburban Hospital, or Children s National Medical Center (CNMC). We will recruit subjects of the Washington Adult Congenital Heart program at CNMC to participate in this study.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Hypothesize that myocardial ischemia, as detectable by quantitative stress perfusion MRI, will predict systolic and diastolic dysfunction in subjects with single ventricle physiology and systemic right ventricles. | 5 years
  The specific aim of this study is to understand whether clinical subendocardial perfusion defects contribute to the late decompensation of adult subjects that have single ventricle physiology and adult subjects that have a systemic right ventricle.

SECONDARY OUTCOMES:
A portion of ventricular systolic or diastolic dysfunction will be predictable based on myocardial fibrosis or scarring related to the underlying pathophysiology of single ventricle physiology & systemic right ventricles or post-surgical... | 5 years
  A portion of ventricular systolic or diastolic dysfunction will be predictable based on myocardial fibrosis or scarring related to the underlying pathophysiology of single ventricle physiology & systemic right ventricles or post-surgical consequences.
myocardial scarring/fibrosis will correlate with symptoms, NYHA functional class and BNP. | 5 years
  myocardial scarring/fibrosis will correlate with symptoms, NYHA functional class and BNP.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Sirajuddin, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (3):
- United States (3):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Verheugt CL, Uiterwaal CS, van der Velde ET, Meijboom FJ, Pieper PG, van Dijk AP, Vliegen HW, Grobbee DE, Mulder BJ. Mortality in adult congenital heart disease. Eur Heart J. 2010 May;31(10):1220-9. doi: 10.1093/eurheartj/ehq032. Epub 2010 Mar 5. PMID 20207625
- [Background] Rutledge JM, Nihill MR, Fraser CD, Smith OE, McMahon CJ, Bezold LI. Outcome of 121 patients with congenitally corrected transposition of the great arteries. Pediatr Cardiol. 2002 Mar-Apr;23(2):137-45. doi: 10.1007/s00246-001-0037-8. Epub 2002 Feb 19. PMID 11889523
- [Background] Meijboom F, Szatmari A, Deckers JW, Utens EM, Roelandt JR, Bos E, Hess J. Long-term follow-up (10 to 17 years) after Mustard repair for transposition of the great arteries. J Thorac Cardiovasc Surg. 1996 Jun;111(6):1158-68. doi: 10.1016/s0022-5223(96)70217-9. PMID 8642816
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-H-0158.html